CLINICAL TRIAL: NCT03716661
Title: Operative vs. Conservative Treatment of Distal Radius Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-10-72-420-17
Record Dates: First submitted 2018-10-05; First posted 2018-10-23 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-05

CONDITIONS: Radius Distal Fracture; Distal Radius Fracture; Radius Fracture Distal
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Arm 1/control group: Participants who are treated with conservative plaster following National Clinical Guidelines.
- Conservative (No Intervention): Arm 2 and 3 consist of participants fulfilling the criteria for operative treatment following National Clinical Guidelines.
  Arm 2: Patients randomized to conservative plaster treatment
- Operative (Other): Arm 2 and 3 consist of participants fulfilling the criteria for operative treatment following National Clinical Guidelines.
  Arm 3: Patients randomized to operative treatment (ORIF)
  Interventions: Procedure: ORIF

INTERVENTIONS:
Procedure: ORIF — Open Reduction Internal Fixation
  Arms: Operative

SUMMARY:
Even though broken wrists are of frequent occurrence, the investigators see a lack of extensive and well executed international studies to clarify which is the best treatment for elderly participants at 65+ years. The Danish Health and Medicines Authority recommend that broken wrists are treated with surgery by using plates and screws when certain radiological criteria are met. Recent studies show that, apparently, there are no advantages by operating rather than treating with plaster when comparing the functional results after one year. However, there is a 30 % risk of serious complications occurring after surgery. This study will examine the pros and cons that participants at 65+ years with broken wrists experience after, by lot, having been treated with either surgery (using plates and screws) or without surgery (using plaster for 5 weeks). The purpose of this study is to compare the complications and level of functioning between participants treated with surgery and without surgery.

ELIGIBILITY:
Inclusion Criteria:

* Danish National Guidelines for operative treatment of distal radius fractures

Exclusion Criteria:

* Patients treated with plaster in Arm1/control group who unexpectedly requires surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related complications at baseline | Baseline
Change in number of participants with treatment-related complications from baseline at week 2 | Week 2
Change in number of participants with treatment-related complications from baseline at week 5 | Week 5
Change in number of participants with treatment-related complications from baseline at month 6 | Month 6
Change in number of participants with treatment-related complications from baseline at 1 year | 1 Year
Range of motion of the wrist at week 5 | Week 5
  a. Flexion (0-90 degrees) b. Extension (0-75 degrees) c. Pronation (0-90 degrees) d. Supination (0-90 degrees) e. Radial flexion (0-25 degrees) f. Ulnar flexion (0-50 degrees)
Change in range of motion of the wrist from week 5 at month 6 | Month 6
  a. Flexion (0-90 degrees) b. Extension (0-75 degrees) c. Pronation (0-90 degrees) d. Supination (0-90 degrees) e. Radial flexion (0-25 degrees) f. Ulnar flexion (0-50 degrees)
Change in range of motion of the wrist from month 6 at 1 year | 1 Year
  a. Flexion (0-90 degrees) b. Extension (0-75 degrees) c. Pronation (0-90 degrees) d. Supination (0-90 degrees) e. Radial flexion (0-25 degrees) f. Ulnar flexion (0-50 degrees)
Level of functioning at baseline | Baseline
  Using QuickDASH (Quick Disabilities of the Arm, Shoulder, and Hand)
Change in level of functioning from baseline at week 2 | Week 2
  Using QuickDASH (Quick Disabilities of the Arm, Shoulder, and Hand)
Change in level of functioning from baseline at week 5 | Week 5
  Using QuickDASH (Quick Disabilities of the Arm, Shoulder, and Hand)
Change in level of functioning from baseline at month 6 | Month 6
  Using QuickDASH (Quick Disabilities of the Arm, Shoulder, and Hand)
Change in level of functioning from baseline at 1 year | 1 Year
  Using QuickDASH (Quick Disabilities of the Arm, Shoulder, and Hand)

CONTACTS AND LOCATIONS:
Locations (1):
- Regionshospitalet Randers, Randers, Denmark

REFERENCES:
- [Derived] Thorninger R, Waever D, Tjornild M, Lind M, Rolfing JD. Prospective Evaluation of Two Cohorts of Non-Operatively Treated Patients with Displaced vs. Minimally and Non-Displaced Distal Radius Fractures. J Clin Med. 2023 Mar 6;12(5):2076. doi: 10.3390/jcm12052076. PMID 36902861
- [Derived] Thorninger R, Waever D, Tjornild M, Lind M, Rolfing JD. VOLCON: a randomized controlled trial investigating complications and functional outcome of volar plating vs casting of unstable distal radius fractures in patients older than 65 years. J Orthop Traumatol. 2022 Nov 28;23(1):54. doi: 10.1186/s10195-022-00673-4. PMID 36443579
- [Derived] Pedersen J, Mortensen SO, Rolfing JD, Thorninger R. A protocol for a single-center, single-blinded randomized-controlled trial investigating volar plating versus conservative treatment of unstable distal radius fractures in patients older than 65 years. BMC Musculoskelet Disord. 2019 Jun 29;20(1):309. doi: 10.1186/s12891-019-2677-y. PMID 31253145